CLINICAL TRIAL: NCT01226225
Title: A Multicentre Trial on the Effectiveness of Physical Rehabilitation of Patients With Coronary Artery Disease: Aerobic Interval Training Versus Moderate Continuous Training.
Acronym: SAINTEX-CAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: KU Leuven (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Antwerp University Hospital, Belgium, Antwerp University Hospital, Belgium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IWT-090870
Record Dates: First submitted 2010-08-19; First posted 2010-10-22 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-08

CONDITIONS: Coronary Artery Disease (CAD);; Myocardial Infarction (MI); Percutaneous Coronary Intervention (PCI); Coronary Artery Bypass Grafting (CABG)
Keywords: Patients with recent coronary event
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic interval training (Experimental)
  Interventions: Behavioral: Aerobic interval training
- Moderate endurance training (Active Comparator)
  Interventions: Behavioral: Moderate endurance training

INTERVENTIONS:
Behavioral: Aerobic interval training — Patients will enter a training program during which aerobic interval training is implemented. Three sessions per week, each lasting for 60 minutes. Total duration of the program: 3 months.
  Arms: Aerobic interval training
Behavioral: Moderate endurance training — Patients will enter a training program during which moderate endurance training is implemented. Three sessions per week, each lasting for 60 minutes. Total duration of the program: 3 months.
  Arms: Moderate endurance training

SUMMARY:
Cardiac rehabilitation, including physical training, has become accepted treatment following myocardial infarction, coronary stent implantation and coronary bypass operation. Besides modifying patients' risk profile for future coronary problems, the focus is on improving exercise capacity. The ability to be able to perform at a higher maximal level is a strong predictor for outcome (new cardiovascular events and mortality). The main purpose of this study is to evaluate whether aerobic interval training outweighs more classical moderate endurance training in improving exercise capacity. During interval training, patients perform exercise at high intensity, but for only a couple of minutes and then recover at a lower intensity. Such intervals are repeated. Preliminary evidence from smaller studies suggests that this type of training leads to a larger increase in exercise capacity, compared to the more traditional endurance training at moderate intensity.

In addition, mechanisms that might explain how this improvement is achieved, as well as safety and impact on quality of life will be studied.

ELIGIBILITY:
Inclusion Criteria:

* patients with CAD (post-PCI, post-MI, post-CABG) and a left ventricular ejection fraction (LVEF) > 40%
* the presence of CAD is defined as prior angiographically documented stenotic lesion(s) of > 75%, or documented myocardial infarction (biochemical, ECG, echocardiographic documentation).
* patients are on optimal medical treatment and stable with regard to symptoms and pharmacotherapy for at least 4 weeks
* in practice, patients will have been hospitalized at least 4 weeks prior to participation in the training programme because of PCI, MI or CABG

Exclusion Criteria:

* significant intercurrent illness last 6 weeks
* known severe ventricular arrhythmia with functional or prognostic significance
* significant myocardial ischemia, hemodynamic deterioration or exercise-induced arrhythmia at baseline testing
* recent CABG (< 30 days)
* other heart disease that limits exercise tolerance (valve disease with significant hemodynamic consequences, hypertrophic cardiomyopathy etc.)
* co-morbidity that may significantly influence one-year prognosis
* functional or mental disability that may limit exercise
* a habit of regular vigorous exercise or participation in a programme of exercise training less than 3 months before inclusion
* acute or chronic inflammatory diseases or malignancy, the use of anti-inflammatory drugs or immune suppression
* glomerular filtration rate (GFR) <25ml/min/1.73m2
* hemoglobin < 10g/dl
* severe chronic obstructive pulmonary disease
* participation in another clinical trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Maximal aerobic capacity, measured during symptom-limited cardio-pulmonary exercise testing | 6 weeks
  Comparison of evolution of maximal aerobic capacity from baseline to 6 weeks
Maximal aerobic capacity, measured during symptom-limited cardio-pulmonary exercise testing | 12 weeks
  Comparison of evolution of maximal aerobic capacity from baseline to 12 weeks
Maximal aerobic capacity, measured during symptom-limited cardio-pulmonary exercise testing | 12 months
  Comparison of evolution of maximal aerobic capacity, measured during symptom-limited cardio-pulmonary exercise testing

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Dienst Cardiale Revalidatie, Cardiologie, Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Leuven, Dienst Hart- en Vaatziekten, Cardiale Revalidatie Herestraat 49, Leuven